CLINICAL TRIAL: NCT04420169
Title: Uniform Communication by Midwives in Preparation for an IVF Treatment
Acronym: UNCOVeR
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201627388
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Communication; IVF
MeSH Terms: conditions — Communication | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRE implementation communication protocol
  Interventions: Other: Questionnaire
- POST implementation communication protocol
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A digital questionnaire to evaluate the communication by midwives will be send out to IVF patients

SUMMARY:
Dutch-speaking women who are about to start an IVF treatment will be approached. If they are willing to participate in the study, they will receive an email with a link to an online questionnaire. This questionnaire will evaluate the communication by the midwive in preparation for an IVF treatment. When 50 women have completed the questionnaire a standardized communication protocol will be enrolled. Once all midwives are trained, 50 other IVF patients will be asked to complete the slightly adapted post questionnaire.The data from both questionnaires will be compared.

ELIGIBILITY:
Inclusion Criteria:

* women who are about to start an IVF treatment at our department

Exclusion Criteria:

* non-Dutch speaking
* women who are counseled by one of the midwives involved in the design of this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Dutch-speaking women who are about to start an IVF treatment at our department.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
How do patients evaluate the communication by the midwife in anticipation of the IVF treatment cycle? | About 20 weeks counting from the launch of each questionnaire or earlier if the target of 50 patients is reached sooner
  Self created questionnaire (no scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No